CLINICAL TRIAL: NCT06622109
Title: PREVENAR 20 SUSPENSION LIQUID FOR INJECTION SPECIAL INVESTIGATION - Investigation in Infants Starting Vaccination at the Age of 2 Month, Inclusive, to 7 Months, Exclusive -
Brief Title: A Study to Learn About the Safety of PREVENAR 20 Vaccine in Infants Aged Between Two to Six Months
Status: Active, not recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7471035; NCT06622109 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-09-28; First posted 2024-10-01 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 20-valent Pneumococcal Conjugate Vaccine: Infants aged 2 months, inclusive to 7 months, exclusive who have been vaccinated with PREVENAR 20 for the first time.
  Interventions: Biological: 20-valent Pneumococcal Conjugate Vaccine

INTERVENTIONS:
Biological: 20-valent Pneumococcal Conjugate Vaccine — Injection in the muscle or subcutaneous , 1 dose 0.5mL

SUMMARY:
The purpose of this study is to learn about the safety of 20-valent Pneumococcal Conjugate Vaccine (PREVENAR 20) under actual clinical practice in Japan.

This study is seeking for infants aged between two months to six months who are vaccinated with PREVENAR 20 for the first time.

Infants aged between two months and six months are normally given four vaccinations. The first three vaccinations are called primary vaccinations and are given with an interval of one month between each vaccination. The fourth vaccination is called the booster and is given between 12 and 15 months of age.

Participants will take part in this study from the day of first vaccination to 28 days after fourth vaccination.

The side effects observed in the participants will be recorded and looked into.

ELIGIBILITY:
Inclusion Criteria:

1. Infants aged 2 months, inclusive, to 7 months, exclusive
2. Those without a history of pneumococcal vaccination including PREVENAR 20
3. Those who are expected to receive 4 doses
4. Those whose parent or legal guardian understands the details of the study and provides consent to provision of information collected in the study to third parties and use of the information for other purposes.

Exclusion Criteria:There are no exclusion criteria for this study.

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants aged 2 months, inclusive, to 7 months, exclusive who PREVENAR 20 for the first time.
Sampling Method: Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Reporting Adverse Reactions(ADRs) | From the first day of each vaccination (1st-4th) up to 28 days after each vaccination (1st-4th).
Percentage of Participants Reporting Serious Adverse Reactions (SADRs) | From the first day of 1st vaccination up to 28 days after 4th vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471035